CLINICAL TRIAL: NCT04898062
Title: Randomized, Controlled, Proof-Of-Concept Trial of CRP-Apheresis for Attenuation of Pulmonary MYocardial and/or Kidney Injury in COvid-19
Brief Title: CRP-Apheresis for Attenuation of Pulmonary, MYocardial and/or Kidney Injury in COvid-19
Acronym: CAPMYKCO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sufficient recruitment of study patients based on the existing inclusion and exclusion criteria is not possible within a reasonable period of time
Sponsor: Pentracor GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-10018-BO
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-09

CONDITIONS: Covid19
Keywords: CRP-apheresis; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRP-apheresis (Active Comparator): Patients randomized to this group will undergo apheresis treatments with treatments every 24 ± 12 h each lasting 4-7 hours, until the CRP value does not rise to ≥ 30 mg/l within 96 h after the last treatment
  Interventions: Device: CRP-apheresis
- Control (No Intervention): Patients randomized to this group will not undergo a apheresis treatments. They will be treated according to the current conventional treatment concept for covid-19 disease

INTERVENTIONS:
Device: CRP-apheresis — The major advantages of depleting C-reactive protein by therapeutic apheresis are the selective removal of the damaging agent by the highly specific ligand and the good controllability of the procedure, since the plasma can be passed over the column as often as necessary to achieve the desired reduction. In addition, treatment can be interrupted or discontinued at any time.
  Other Names: CRP-depletion
  Arms: CRP-apheresis

SUMMARY:
The 'CAPMYKCO' study is a randomized controlled, open-label, single center proof of concept trial. The aim of this study is to evaluate whether a CRP-apheresis in addition to the current standard therapy is intended to mitigate the severity of the disease course of SARS-CoV-2, especially with regard to tissue injury in the lungs, heart and kidneys and their consequences.

CRP-apheresis should reduce the necessity and duration of non-invasive/invasive ventilation requirements compared to the control group.

The influence of CRP-apheresis on the attenuation of pulmonary, myocardial and/or kidney tissue injury as well as the course of the COVID-19 disease will also be demonstrated by evaluating various biomarkers, several clinical scoring systems, and the duration of intensive care medical treatment.

DETAILED DESCRIPTION:
The prognostic value of C-reactive protein (CRP) in assessing disease progression in COVID-19 is well known: The steeper the CRP rise in the days after infection and the higher the CRP concentration at hospitalization, the worse the prognosis. It is believed that CRP concentration not only reflects tissue damage but also causally contributes to the severity of the damage that occurs. CRP apheresis effectively limits CRP rise, which may lead to improved prognosis. CRP apheresis is a therapeutic hemapheresis procedure that selectively removes C-reactive protein from the patient's plasma. Other causal therapies for immediate selective reduction of CRP in the acute phase of disease are not currently available.

In the planned 'CAPMYKCO' study, CRP-apheresis in addition to current standard COVID-19 therapy is expected to mitigate the severity of disease progression, particularly with regard to tissue injury in the lungs, the heart and/or the kidneys and their respective clinical consequences.

CRP-apheresis treatment in COVID-19 patients should reduce the necessity and duration of non-invasive / invasive ventilation compared to the control group.

The influence of CRP-apheresis on the course of the COVID-19 disease will also be demonstrated by evaluating different organ biomarkers and the duration of intensive medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS CoV-2 infection (PCR-test)
* Oxygen therapy (maximum 'high-flow' therapy)
* CRP plasma concentration ≥ 50 mg/l and/or
* CRP increase ≥ 15 mg/l within 24 h after admission.
* Completed informed consent and written informed consent.
* Legal capacity

Exclusion Criteria:

* Age < 18 years
* Pregnancy / lactation period
* Invasive, mechanical ventilation
* Extracorporeal membrane oxygenation (ECMO)
* Participation in other interventional trials
* Extracorporeal membrane oxygenation (ECMO) support
* Participation in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Necessity and duration of non-invasive/ invasive ventilation | through study completion, an average of 14 days
  In the intervention group, a reduced necessity and duration of non-invasive/ invasive ventilation is expected.

SECONDARY OUTCOMES:
Length of intensive care unit stay | through study completion, an average of 14 days
  In the intervention group, a shorter intensive care unit stay is expected.
Necessity of endotracheal intubation | through study completion, an average of 14 days
  In the intervention group, a reduced necessity of endotracheal intubation is expected.
Reduction of lung injury | through study completion, an average of 14 days
  In the intervention group, a reduced lung injury as reflected by peripheral oxygen saturation, oxygen supplementation, Horovitz index, lung injury score is expected.
Reduction of myocardial damage | up to 10 days
  In the intervention group, a reduced myocardial damage as reflected by hs troponin, creatin kinase, creatin kinase MB fraction is expected.
Reduction of kidney damage | up to 10 days
  In the intervention group, a reduced kidney damage as reflected by creatinine, glomerular filtration rate, onset of dialysis, CKD stadium is expected.
Improvement in general immune status | up to 10 days
  In the intervention group, an improved general immune status as reflected by CRP, fibrinogen, leukocytes, thrombocytes and lactate dehydrogenase is expected.
Cardiovascular, respiratory and renal SOFA score | through study completion, an average of 14 days
  In the intervention group, improvements in cardiovascular, respiratory and renal SOFA scores are expected.
  *(Vincent JL: The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. In:Intensive Care Med 1996:22;707-10.)
Respiratory events | through study completion, an average of 14 days
  In the intervention group, a reduction of respiratory events (pulmonary embolism) is expected.
Myocardial events | through study completion, an average of 14 days
  In the intervention group, a reduction of cardial events (cardiac arrhythmias, myocardial infarction, cardiopulmonary resuscitation, low cardiac output syndrome (LCOS), operation, percutaneous coronary intervention (PCI), angina pectoris) is expected.
Renal events | through study completion, an average of 14 days
  In the intervention group, a reduction of renal events (onset of dialysis requirement, deterioration of renal function (CKD increase) is expected.
Safety of CRF apheresis | through study completion, an average of 14 days
  In the intervention group, the absence of serious incidents is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Thielmann, Prof., Principal Investigator — West-German Heart and Vascular Center, University Duisburg-Essen
Locations (4):
- Germany (4):
  - West-German Heart and Vascular Center, University Duisburg-Essen, Essen, North Rhine-Westphalia
  - Gemeinschaftskrankenhaus Havelhöhe gGmbH, Berlin
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikverbund Allgäu gGmbH, Kempten

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueller AA, Tamura T, Crowley CP, DeGrado JR, Haider H, Jezmir JL, Keras G, Penn EH, Massaro AF, Kim EY. Inflammatory Biomarker Trends Predict Respiratory Decline in COVID-19 Patients. Cell Rep Med. 2020 Nov 17;1(8):100144. doi: 10.1016/j.xcrm.2020.100144. Epub 2020 Oct 29. PMID 33163981
- [Background] Smilowitz NR, Kunichoff D, Garshick M, Shah B, Pillinger M, Hochman JS, Berger JS. C-reactive protein and clinical outcomes in patients with COVID-19. Eur Heart J. 2021 Jun 14;42(23):2270-2279. doi: 10.1093/eurheartj/ehaa1103. PMID 33448289
- [Background] Kunze R. C-Reactive Protein: From Biomarker to Trigger of Cell Death? Ther Apher Dial. 2019 Dec;23(6):494-496. doi: 10.1111/1744-9987.12802. No abstract available. PMID 31788974
- [Background] Torzewski J, Heigl F, Zimmermann O, Wagner F, Schumann C, Hettich R, Bock C, Kayser S, Sheriff A. First-in-Man: Case Report of Selective C-Reactive Protein Apheresis in a Patient with SARS-CoV-2 Infection. Am J Case Rep. 2020 Jul 14;21:e925020. doi: 10.12659/AJCR.925020. PMID 32661220
- [Background] Pepys MB. C-reactive protein predicts outcome in COVID-19: is it also a therapeutic target? Eur Heart J. 2021 Jun 14;42(23):2280-2283. doi: 10.1093/eurheartj/ehab169. No abstract available. PMID 33778886
- [Background] Murray JF, Matthay MA, Luce JM, Flick MR. An expanded definition of the adult respiratory distress syndrome. Am Rev Respir Dis. 1988 Sep;138(3):720-3. doi: 10.1164/ajrccm/138.3.720. No abstract available. PMID 3202424
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Ringel J, Ramlow A, Bock C, Sheriff A. Case Report: C-Reactive Protein Apheresis in a Patient With COVID-19 and Fulminant CRP Increase. Front Immunol. 2021 Aug 2;12:708101. doi: 10.3389/fimmu.2021.708101. eCollection 2021. PMID 34408751
- [Background] Torzewski J, Zimmermann O, Kayser S, Heigl F, Wagner F, Sheriff A, Schumann C. Successful Treatment of a 39-Year-Old COVID-19 Patient with Respiratory Failure by Selective C-Reactive Protein Apheresis. Am J Case Rep. 2021 Aug 5;22:e932964. doi: 10.12659/AJCR.932964. PMID 34351878
- [Background] Schumann C, Heigl F, Rohrbach IJ, Sheriff A, Wagner L, Wagner F, Torzewski J. A Report on the First 7 Sequential Patients Treated Within the C-Reactive Protein Apheresis in COVID (CACOV) Registry. Am J Case Rep. 2022 Jan 10;23:e935263. doi: 10.12659/AJCR.935263. PMID 35007274